CLINICAL TRIAL: NCT04784325
Title: AMH^2: Anti-Müllerian Hormone - At My Home
Brief Title: Anti-Mullerian Hormone - At My Home
Acronym: AMH^2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turtle Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 009
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Fertility Risk

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women recruited from a general population subject to I/E criteria (Experimental): All study participants will administer three blood collection modalities (2 TAP II, 1 ADx card, and phlebotomist-performed venipuncture).
  Interventions: Diagnostic Test: Blood draw through TAP II; Diagnostic Test: Blood draw through ADx cardT; Diagnostic Test: Blood draw through standard venipuncture

INTERVENTIONS:
Diagnostic Test: Blood draw through TAP II — Two self-administered blood draws through TAP II device
Diagnostic Test: Blood draw through ADx cardT — One self-administered ADx card blood draw
Diagnostic Test: Blood draw through standard venipuncture — One phlebotomist-performed standard venipuncture

SUMMARY:
The AMH^2 (Anti-Mullerian Hormone - At My Home) study is a head-to-head-to-head validation study aiming to evaluate the concordance of AMH levels found in blood collected via three different routes: collected at-home using the TAP II device, drawn through standard venipuncture techniques, and collected with the ADx card, another at-home collection device widely available on the market for commercial use.

DETAILED DESCRIPTION:
Today, information regarding fertility potential is challenging to obtain for healthy women; clinically meaningful in-clinic testing is limited by physician availability and patient willingness to undergo testing in-clinic. Meanwhile, at-home hormonal bloodwork relies on the use of an ADx card, and is not widely accepted as clinically reliable by the medical community. The Sponsor is developing a comprehensive home fertility assessment to enable couples to proactively estimate and manage their fertility and family building options. Accurate and reliable at-home AMH testing is necessary to reach this goal.

This study aims to validate the clinical excellence and medical accuracy of blood drawn via the TAP II device relative to a standard in-clinic venipuncture draw and other options available on the market to support emerging telemedicine care models. In doing so, the Sponsor may receive CLIA validation for the TAP II in AMH testing and commercialize a Lab Developed Test.

ELIGIBILITY:
Study Participants

Inclusion Criteria:

* Women between the ages of 20 and 39, inclusive (two age brackets above)
* Women able to freely give consent electronically, given COVID. For the purposes of this study, this is defined as women who speak native or fluent English; and have a high school degree or equivalent, and who are otherwise, in the professional judgement of the PI, able to give informed consent
* Women who are in driving distance from Boston

Exclusion Criteria:

* Turtle Health employees
* Women who do not speak English natively or fluently
* Women who have recently given birth, and have had fewer than 3 postpartum menstrual cycles
* Women who have recently had a stillbirth or abortion more than 20 weeks (subject to the 3 postpartum menstrual cycles above). Miscarriages or abortions less than 20 weeks are subject to wait 2 cycles
* Women who are currently pregnant or may be pregnant
* Women who have known blood hypo- or hypercoagulability disorders or known blood clotting issues
* Any woman the PI believes is not capable of giving independent, informed consent

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation (r-squared) of the AMH levels resulting from the shipped TAP II samples and venipuncture samples. | Lab analysis 72 hours after ADx card/venipuncture/TAP II hand delivery
  Evaluate the concordance of the TAP blood collection device after shipment with in-clinic blood collection for AMH.

SECONDARY OUTCOMES:
Correlation (r-squared) of AMH levels from stored TAP II samples and venipuncture samples | Lab analysis 72 hours after ADx card/venipuncture/TAP II hand delivery
  Evaluate the concordance of the TAP blood collection device without shipment with in-clinic blood collection for AMH for control versus venipuncture "ground truth".
Correlation (r-squared) of AMH levels from stored ADx samples and venipuncture samples. | Lab analysis 72 hours after ADx card/venipuncture/TAP II hand delivery
  Evaluate the concordance of the ADx card comparator device with in-clinic blood collection for AMH for control versus venipuncture "ground truth".
Number of women changing risk bands | Lab analysis 72 hours after ADx card/venipuncture/TAP II hand delivery
  The number of participants who move to a different risk strata for their age and hormonal birth control status. This will be defined by changing to a different row for their AMH concentration range, treating venipuncture as the "Gold Standard" and comparing the number of women who move rows utilizing their TAP draws or ADx card draw.
NPS superiority | Survey collected within 3 days of blood draw
  Superiority of net promoter score of TAP II device compared to venipuncture as measured by a post-draw survey (calculated as a standard NPS: 9/10 scores - 0-6 scores).
Self-reported pain | Survey collected within 3 days of blood draw
  Self-reported pain of different draw methods as measured by a post-draw using the Stanford Pain Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anatte E Karmon, Harvard University, Principal Investigator — Fertility Institute of Hawaii
Locations (1):
- Turtle Health Pop-up Clinic, Brookline, Massachusetts, United States

REFERENCES:
- [Derived] Silliman E, Chung EH, Fitzpatrick E, Jolin JA, Brown M, Hotaling J, Styer AK, Karmon AE. Evaluation of at-home serum anti-Mullerian hormone testing: a head-to-head comparison study. Reprod Biol Endocrinol. 2022 Sep 1;20(1):131. doi: 10.1186/s12958-022-01004-2. PMID 36050723